CLINICAL TRIAL: NCT01827319
Title: A Multi-Center Single Arm Observational Registry of the Cardiogenesis Holmium: YAG Laser System Transmyocardial Revascularization for Angina Reduction
Brief Title: Cardiogenesis Transmyocardial Revascularization Registry
Acronym: ANGINA RELIEF
Status: Completed | Type: Observational
Sponsor: Cardiogenesis Corporation, a wholly-owned subsidiary of CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TMR1201.001-M
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Class IV Angina
Keywords: Angina; Transmyocardial revascularization
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of the registry are as follows:

* Track "real world" performance outcomes and physician experience using the Cardiogenesis Laser System;
* Further define the disease characteristics of the population being treated;
* Examine transmyocardial revascularization (TMR) usage characteristics and 30-day outcomes;
* Further assess the 30-day postoperative risk factors for adverse events. To limit the potential for bias, all patients eligible for TMR treatment who meet the Inclusion and Exclusion Criteria are to be offered the opportunity to enroll in the study at participating centers.

DETAILED DESCRIPTION:
The objectives of this patient registry, which collects data on the Cardiogenesis Laser System, include: provide further information on the disease characteristics of the population being treated, examine TMR usage characteristics, monitor 30-day postoperative mortality and MACE rates, and assess preoperative and operative risk factors for adverse events.

To limit the potential for bias, all patients eligible for TMR treatment who meet the Inclusion and Exclusion Criteria are to be offered the opportunity to enroll in the study at participating centers. Patient consent indicates approval to allow collection of their confidential data; nonetheless, their identity will not be disclosed in any publication of this study.

The primary endpoint to be assessed in this study is:

• All-cause 30-day mortality

Additional endpoints to be assessed in this study are:

• Major adverse cardiovascular events (MACE) rate, defined as the incidence of cardiac-related death, myocardial infarction (Q-wave and non Q-wave), congestive heart failure, cerebrovascular accident, and serious arrhythmia in the 30-day postoperative period.

The definitions for these events are as follows:

Cardiac-related death: any death that is not clearly attributable to a non-cardiac cause and includes death due to any of the following: acute myocardial infarction, heart failure, cardiogenic shock, pulmonary edema, cardiac tamponade, arrhythmia, or post-procedural complications (i.e., bleeding).

Q-wave myocardial infarction: the appearance of new Q waves of 40 or more milliseconds in 2 or more contiguous leads and elevation of CK-MB.

Non Q-wave myocardial infarction: the elevation of total CK more than twice normal with elevated CK-MB.

Congestive heart failure: Symptoms of pulmonary vascular congestion or a low output state that is due to left ventricular failure and is new in onset or results in re-hospitalization.

Cerebrovascular accident: Any sudden development of neurological deficits due to vascular lesions of the brain such as hemorrhage, embolism, or thrombosis that persists for > 24 hours.

Serious arrhythmia: Supraventricular or ventricular arrhythmias that require sustained intravenous pharmacologic treatment, temporary or permanent pacing, or immediate electrical cardioversion or defibrillation. Arrhythmias resulting in syncope, myocardial ischemia, or death are also classified as serious.

Any other serious operative complications related to the procedure: example: major bleeding requiring transfusion.

Each contributing site is required to complete the Enrollment Failure Log Form for all patients undergoing TMR, but not enrolled into the registry due to inclusion/exclusion criteria failure or did not consent for registry participation. If the decision to perform TMR is done intra-operatively, the patient will be approached for participation in the registry after the procedure. No data should be collected prior to patient consent to take part in the registry.

All data collected must be supported by source documents found at the site. Patient medical records, hospital charts, operative reports, laboratory and diagnostic testing results, office visits, source document worksheets as supplied by the Sponsor, etc. will be utilized for collection of relevant data. All data is subject to 100% source document review by Sponsor personnel and/or a representative of the Sponsor at Sponsor's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Class IV angina (according to Canadian Cardiovascular Society Angina Scale)
* Patients with regions of myocardium in the distal two-thirds of the left ventricle with reversible ischemia and who are not eligible for direct coronary revascularization (e.g., CABG or PTCA)

Exclusion Criteria:

* Age less than18 years
* Severely unstable angina (un-weanable from intravenous anti-anginals for 48-hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the eligibility criteria and undergo TMR at the selected centers will be provided an opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Capps, MS, Study Director — CryoLife, Inc.
Locations (24):
- United States (24):
  - University of Arizona, Tuscon, Arizona
  - California Cardiac Surgeons, Bakersfield, California
  - The Vo Group, Fountain Valley, California
  - Hurwitz & Roberts Med Corp, Glendale, California
  - Advanced Cardiothoracic Surgery Medical Group, Los Angeles, California
  - Soltero & Yasuda Associates Cardiothoracic & Vascular Medical Group, Northridge, California
  - Cardiovascular & Thoracic Surgeons of Ventura County, APC, Oxnard, California
  - Joseph W. Wilson, MD, Inc., Rancho Mirage, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Cardiothoracic and Vascular Surgical Associates, Jacksonville, Florida
  - Coastal Cardiovascular and Thoracic Associates, PA, Ormond Beach, Florida
  - Georgia Health Sciences University Research Institute, Inc., Augusta, Georgia
  - Lexington Cardiac Research Foundation, Inc., Lexington, Kentucky
  - Owensboro Health, Inc., Owensboro, Kentucky
  - Regional Heart & Lung Surgery, Paducah, Kentucky
  - Saint Luke's Hospital, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Feinstein Institute for Medical Research, New York, New York
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - East Tennessee Cardiovascular Surgery Group, Knoxville, Tennessee
  - Tristar Cardiovascular Surgery, Nashville, Tennessee
  - Cardiopulmonary Research Science and Technology Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Received TMR and Enrolled in ANGINA RELIEF Registry
Started | 203
Completed | 200
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Received TMR and Enrolled in ANGINA RELIEF Registry
Number analyzed (Participants) | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 203

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Description: Number of Participant Deaths
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Received TMR and Enrolled in ANGINA RELIEF Registry
Number analyzed (Participants) | 200
participants | 1

2. Secondary Outcome: Major Adverse Cardiovascular Events (MACE) Rate, Defined as the Incidence of Cardiac-related Death, Myocardial Infarction (Q-wave and Non Q-wave), Congestive Heart Failure, Cerebrovascular Accident, and Serious Arrhythmia
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Received TMR and Enrolled in ANGINA RELIEF Registry
Number analyzed (Participants) | 200
participants | 19

3. Secondary Outcome: 2 CCS Angina Class Reduction
Description: Canadian Cardiovascular Society (CCS) Angina Class-Class I: Ordinary physical activity does not cause angina, such as walking and climbing stairs. Angina with strenuous or rapid or prolonged exertion at work or recreation; Class II: Slight limitation of ordinary activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, or in cold, or in wind, or under emotional stress, or only during the few hours after awakening. Walking more than two blocks on the level and climbing more than one flight of ordinary stairs at a normal pace and in normal conditions; Class III: Marked limitation of ordinary physical activity. Walking one or two blocks on the level and climbing one flight of stairs in normal conditions and at normal pace; Class IV: Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Received TMR and Enrolled in ANGINA RELIEF Registry
Number analyzed (Participants) | 185
participants | 183

ADVERSE EVENTS:
Arm/Group | Received TMR and Enrolled in ANGINA RELIEF Registry
Serious Adverse Events (participants affected / at risk) | 19/200
Other Adverse Events (participants affected / at risk) | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Received TMR and Enrolled in ANGINA RELIEF Registry (N=200)
Major Adverse Cardiac Event (Cardiac disorders) | 19 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Additionally, Sponsor has the right to request removal of any confidential information prior to publication.